CLINICAL TRIAL: NCT02158039
Title: Endoscopic Ultrasound-guided Ethanol Injection of Pancreatic Cystic Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Topazian, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 498-04
Record Dates: First submitted 2013-09-30; First posted 2014-06-06 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms, Cystic, Mucinous, and Serous
Keywords: Intraductal Papillary Mucinous Neoplasm; Mucinous Cystic Neoplasm; Endoscopic Ultrasound; Ethanol
MeSH Terms: conditions — Neoplasms, Cystic, Mucinous, and Serous | interventions — Ethanol; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pancreatic Cyst Ethanol Injection (Experimental): EUS-guided lavage of a pancreatic cyst with ethanol solution. The ethanol solution was diluted to 80% using normal saline. Final solution also contained 1% lidocaine except in patients allergic to local anesthetics. The ethanol solution was injected into pancreatic cysts at a volume equal to 90% of the aspirated cyst volume. In subjects undergoing re-treatment of a cyst, ethanol was diluted to 90% using normal saline, and injected in a volume equal to 100% of the aspirated cyst volume.
  Interventions: Drug: Ethanol; Drug: Lidocaine

INTERVENTIONS:
Drug: Ethanol — EUS-guided lavage of a pancreatic cystic neoplasm with ethanol solution. Ethanol was diluted to 80% using normal saline.
Drug: Lidocaine — The final solution contained 1% lidocaine except in subjects allergic to local anesthetics.

SUMMARY:
Cystic tumors of the pancreas are fluid-filled growths. They are often treated by surgical removal. A safe and effective non-surgical treatment is desirable. Ethanol (alcohol) injection may treat cysts by killing the lining cells of the cyst, and is an accepted treatment for cysts of other organs. In this study, participants with pancreatic cysts underwent endoscopic ultrasound (EUS) guided ethanol injection of pancreatic cysts. This was a pilot study to assess safety and efficacy.

The hypotheses of this study were 1) complications of EUS guided ethanol injection requiring hospitalization will occur in <10% of subjects, and 2) EUS guided ethanol injection, with retreatment as necessary, will ablate at least 50% of pancreatic cysts.

DETAILED DESCRIPTION:
EUS is performed via the mouth under sedation. After a needle is placed into the pancreas cyst under EUS guidance, an ethanol solution is placed into the cyst via the needle. The ethanol solution is withdrawn and new ethanol injected, and this process is continued for 5 minutes, repeatedly washing the cyst with the ethanol solution.

After this treatment, usual clinical follow-up is obtained including assessments of the cyst by CT or MRI scans. If a cyst of significant size persists, additional EUS-guided ethanol injections of the cyst were offered.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a pancreatic cystic lesion, > 1 cm in maximum diameter
2. Treatment of the cystic lesion is desired due to symptoms or concern for subsequent malignancy
3. Age > or = 18 years
4. Able to give informed consent
5. Surgical treatment has been considered, and a surgical consultation offered to the patient, but:

   1. Subject's cyst does not meet consensus criteria for surgical resection, or
   2. Subject is deemed a poor operative candidate, or
   3. Ethanol ablation would allow a subtotal rather than total pancreatectomy, or
   4. Subject has decided not to undergo surgical treatment.

Exclusion Criteria:

1. Known or suspected pregnancy, or nursing
2. History of pancreatitis within past 3 months
3. Main pancreatic duct is dilated to > 4mm in neck, body, or tail
4. Cyst is known to communicate with the pancreatic duct
5. Cyst has a primarily microcystic architecture on EUS
6. Cyst is immediately adjacent to the main pancreatic duct on EUS
7. Cyst has a connection to the main pancreatic duct seen during EUS
8. During initial cyst aspiration, more fluid is recovered than expected (suggesting communication to the main pancreatic duct)
9. Pancreatic cytology has demonstrated cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Topazian, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing can be arranged and will require IRB approval

REFERENCES:
- [Background] Gomez V, Takahashi N, Levy MJ, McGee KP, Jones A, Huang Y, Chari ST, Clain JE, Gleeson FC, Pearson RK, Petersen BT, Rajan E, Vege SS, Topazian MD. EUS-guided ethanol lavage does not reliably ablate pancreatic cystic neoplasms (with video). Gastrointest Endosc. 2016 May;83(5):914-20. doi: 10.1016/j.gie.2015.08.069. Epub 2015 Sep 9. PMID 26363331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the Mayo Clinic Pancreas Clinic or the Mayo Clinic Interventional Endoscopy Unit in Rochester, Minnesota between April 2004 and August 2014.
Pre-assignment Details: Thirty-three subjects were enrolled, of whom 23 underwent study procedures and were considered accrued. Of the remaining 10, one withdrew and the other nine were excluded for a variety of per-protocol reasons including cysts found to communicate with pancreatic duct. Study was closed when an interim analysis showed low efficacy.
Groups:
- Pancreatic Cyst Ethanol Injection: Endoscopic ultrasound (EUS)-guided lavage of a pancreatic cyst with ethanol solution. The ethanol solution was diluted to 80% using normal saline. Final solution also contained 1% lidocaine except in patients allergic to local anesthetics. The ethanol solution was injected into pancreatic cysts at a volume equal to 90% of the aspirated cyst volume. In subjects undergoing re-treatment of a cyst, ethanol was diluted to 90% using normal saline, and injected in a volume equal to 100% of the aspirated cyst volume.
Period: Overall Study
Arm/Group | Pancreatic Cyst Ethanol Injection
Started | 33
Completed | 23
Not Completed | 10
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 9

BASELINE CHARACTERISTICS:
Population: Only subjects who received the study intervention, endoscopic ultra sound (EUS)- guided ethanol lavage were included in the baseline analysis.
Arm/Group | Pancreatic Cyst Ethanol Injection
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 70 [53 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events include pancreatitis, bleeding, perforation, any other occurrence resulting in hospitalization, medical treatment, surgery, death, or disability
Time Frame: 1 year after final treatment
Measure: Number; unit: participants
Arm/Group | Pancreatic Cyst Ethanol Injection
Number analyzed (Participants) | 23
participants
  Number of participants with adverse events | 7
  Number of participants without adverse events | 16

2. Primary Outcome: Number of Subjects With Complete or Partial Ablation of the Treated Cyst
Description: Complete or partial ablation of cysts will be defined by the presence of a persistent cystic structure, and its volume and maximum diameter, as determined by cross-sectional imaging studies (CT, MR)
Time Frame: 1 year after final treatment
Measure: Number; unit: participants
Arm/Group | Pancreatic Cyst Ethanol Injection
Number analyzed (Participants) | 23
participants
  Complete ablation of treated cyst | 2
  Greater than or equal to 80% cyst volume reduction | 10
  Less than 80% cyst volume reduction | 10
  Cyst volume increase | 1

ADVERSE EVENTS:
Time Frame: Participants were followed up at 3 days, 6 and 12 months, and then yearly after the last endoscopic ultrasound-guided ethanol lavage procedure, approximately 72 months.
Arm/Group | Pancreatic Cyst Ethanol Injection
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Cyst Ethanol Injection (N=23)
Acute interstitial pancreatitis (Gastrointestinal disorders) | 1 (1) — Required hospitalization
Death due to pancreatic adenocarcinoma (Gastrointestinal disorders) | 1 (1)
Death due to metastatic gallbladder carcinoma (Gastrointestinal disorders) | 1 (1)
Death due to congestive heart failure (Cardiac disorders) | 1 (1)
Death due to biventricular systolic heart failure (Cardiac disorders) | 1 (1)
Death due to motor vehicle accident (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Cyst Ethanol Injection (N=23)
Transient abdominal pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size was small, and a control group was not included. Neither cyst histology not degree of epithelial ablation was assessed by surgical resection in any of the study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes